CLINICAL TRIAL: NCT02286154
Title: Therapeutic Response Evaluation and Adherence Trial (TREAT): A Prospective Study of Hydroxyurea for Children With Sickle Cell Anemia
Brief Title: Therapeutic Response Evaluation and Adherence Trial (TREAT)
Acronym: TREAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC_TREAT
Record Dates: First submitted 2014-10-01; First posted 2014-11-07 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Anemia, Sickle Cell
Keywords: Hydroxyurea; Sickle Cell; Pharmacokinetics; dynamics; genomics
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxyurea (Experimental): All enrolled participants will receive hydroxyurea, but upon enrollment, participants will be identified as part of the "New Cohort" or "Old Cohort" "New Cohort" participants include those who are not receiving hydroxyurea therapy upon study entry. "Old Cohort" participants include those who are already receiving hydroxyurea therapy upon study entry. New Cohort participants will have starting dose predicted using PK/PD data and Old Cohort participants will continue dosing per clinical guidelines.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — For New Cohort participants, PK/PD data will be used to predict the most effective maximum tolerated dose. Old Cohort participants will receive hydroxyurea escalated to MTD as per local clinical guidelines.

SUMMARY:
The primary objectives of this prospective study of hydroxyurea for children with sickle cell anemia are 1) Develop and prospectively evaluate a population pharmacokinetic/pharmacodynamics model to predict the maximum tolerated dose (MTD); 2) Identify urine biomarkers of hydroxyurea adherence using a novel metabolomics approach; 3) Identify pharmacogenomics modifiers of hydroxyurea MTD; and 4) Longitudinal monitoring of the effect of hydroxyurea upon organ function and quality of life.

DETAILED DESCRIPTION:
There is now ample clinical evidence that hydroxyurea is a safe and effective medication for adults and children with sickle cell anemia (SCA), and most hematologists agree the short-term safety and efficacy of hydroxyurea has been proven. The National Heart, Lung, and Blood Institute have recently released evidence-based guidelines for SCA, recommending that hydroxyurea be offered to all affected children as young as nine months of age, regardless of clinical severity. Despite the overwhelming evidence demonstrating safety and efficacy, hydroxyurea remains underutilized for a variety of reasons. In this prospective study, the investigators will utilize innovative strategies designed to address and overcome some of the barriers that currently limit the use of hydroxyurea for children with SCA. The investigators will utilize novel laboratory techniques and pharmacometric modeling in order to accurately predict the most effective hydroxyurea dose referred to as the maximum tolerated dose. The investigators aim to develop a screening urine test to objectively and accurately determine adherence to hydroxyurea therapy. In addition, the study will document critical laboratory and clinical characteristics of this unique population of patients with SCA who begin hydroxyurea at a young age.

This study will follow two groups of patients. The first group, referred to as the New Cohort, will include mostly young infants who are not receiving hydroxyurea therapy upon entering the study. The starting dose of hydroxyurea for each of the participants in the New Cohort will be individually determined using the novel population PK/PD dose-prediction model. The second group of study participants, referred to as the Old Cohort, will include patients who are already receiving hydroxyurea therapy upon study entry. Both the Old and New Cohort (New Cohort) will be included in the development of a urine biomarker of adherence and will be followed throughout the study to document the effect hydroxyurea has upon organ function and quality of life. It is important to note that this is not a therapeutic drug trial. Prior to enrollment in the study, participants, along with their families and clinical providers, have decided to initiate hydroxyurea therapy for clinical indications. Except for the dose prediction model for the New Cohort, participants will be treated and monitored according to the routine clinical practice guidelines of the Cincinnati Children's Hospital Comprehensive Sickle Cell Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell anemia (HbSS or Hbβ0-thalassemia)
2. Age 6 months to 21 years at the time of enrollment
3. Clinical decision by patient, family, and healthcare provider to initiate hydroxyurea therapy, including patients who are transitioning from chronic transfusions to hydroxyurea therapy

Exclusion Criteria:

1. Family unwillingness to sign informed consent or comply with study treatments

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to Reach Maximum Tolerated Dose (months) | Twelve months
  Time it takes to reach maximum tolerated dose (MTD) of hydroxyurea quantified in months.

SECONDARY OUTCOMES:
Hydroxyurea adherence | Monthly until MTD then yearly up to ten years
  Hydroxyurea adherence as measured by analysis of urine metabolites
Neurological function | Yearly
  Neurological function as measured by transcranial Doppler study (yearly), brain MRI (every 5 years beginning at age 5).
Non-invasive Transcranial Cerebral Oximetry | Monthly until MTD then every six months, up to ten years
  Non-invasive transcranial cerebral oximetry
Splenic function | Annually up to ten years
  Splenic function as measured by pocked red blood cell counts ("pit counts")
Kidney function | Annually, up to ten years
  Kidney function as measured by BUN/creatinine, urinalysis, and cystatin-C
Cardiac function (assessment and growth) | Every Five Years, up to 21 years of age
  Cardiac function as measured by echocardiogram and ECG
Assessment of Growth | Every six months, up to ten years
  Assessment of growth as defined by height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Charles Quinn, MD, MS, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Power-Hays A, McElhinney KE, Williams TN, Mochamah G, Olupot-Olupot P, Paasi G, Reid ME, Rankine-Mullings AE, Opoka RO, John CC, McGann PT, Quinn CT, Punt NC, Smart LR, Stuber SE, Latham TS, Vinks AA, Ware RE. Hydroxyurea pharmacokinetics in children with sickle cell anemia across different global populations. Blood Adv. 2026 Jan 27;10(2):418-427. doi: 10.1182/bloodadvances.2025017254. PMID 41026975
- [Derived] Quinn CT, Niss O, Dong M, Pfeiffer A, Korpik J, Reynaud M, Bonar H, Kalfa TA, Smart LR, Malik P, Ware RE, Vinks AA, McGann PT. Early initiation of hydroxyurea (hydroxycarbamide) using individualised, pharmacokinetics-guided dosing can produce sustained and nearly pancellular expression of fetal haemoglobin in children with sickle cell anaemia. Br J Haematol. 2021 Aug;194(3):617-625. doi: 10.1111/bjh.17663. Epub 2021 Jul 5. PMID 34227124
- [Derived] Sadaf A, Quinn CT, Korpik JB, Pfeiffer A, Reynaud M, Niss O, Malik P, Ware RE, Kalfa TA, McGann PT. Rapid and automated quantitation of dense red blood cells: A robust biomarker of hydroxyurea treatment response. Blood Cells Mol Dis. 2021 Sep;90:102576. doi: 10.1016/j.bcmd.2021.102576. Epub 2021 May 11. No abstract available. PMID 34020272
- [Derived] McGann PT, Niss O, Dong M, Marahatta A, Howard TA, Mizuno T, Lane A, Kalfa TA, Malik P, Quinn CT, Ware RE, Vinks AA. Robust clinical and laboratory response to hydroxyurea using pharmacokinetically guided dosing for young children with sickle cell anemia. Am J Hematol. 2019 Aug;94(8):871-879. doi: 10.1002/ajh.25510. Epub 2019 Jun 12. PMID 31106898
- [Derived] Dong M, McGann PT, Mizuno T, Ware RE, Vinks AA. Development of a pharmacokinetic-guided dose individualization strategy for hydroxyurea treatment in children with sickle cell anaemia. Br J Clin Pharmacol. 2016 Apr;81(4):742-52. doi: 10.1111/bcp.12851. Epub 2016 Feb 5. PMID 26615061